CLINICAL TRIAL: NCT05607940
Title: A Multi-center, Single Blinded Randomized Trial Investigating Indications Based Blood Transfusion Practices in Patients With Major Oncological Surgery
Brief Title: Effect of Indication Based Blood Product Transfusion in Patients Undergoing Major Oncological Surgery
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022_XB1028
Record Dates: First submitted 2022-10-28; First posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-10

CONDITIONS: Blood Transfusion
Keywords: blood loss，transfusion，oncological surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- blood volume loss based blood transfusion (Experimental): intraoperative blood transfusion begin once blood volume loss over 400ml
  Interventions: Procedure: blood volume loss based blood transfusion
- hemoglobin concentration based blood transfusion (Active Comparator): intraoperative blood transfusion begin once hemoglobin concentration below 70g/L
  Interventions: Procedure: hemoglobin concentration based blood transfusion

INTERVENTIONS:
Procedure: blood volume loss based blood transfusion — Blood transfusion is indicated based on the estimated intraoperative blood loss. When intraoperative blood loss exceeds 400ml, blood transfusion begin. At the end of the operation, we ensure that the volume of blood transfusion is no greater than the anticipated blood loss.
  Arms: blood volume loss based blood transfusion
Procedure: hemoglobin concentration based blood transfusion — Blood transfusion is indicated based on the intraoperative hemoglobin concentration. Intraoperative blood transfusion begins when hemoglobin concentration is blow 70g/L. Intraoperative blood transfusion stops when hemoglobin concentration reaches 80g/L
  Arms: hemoglobin concentration based blood transfusion

SUMMARY:
Investigators aimed to compare the effect on different indications (blood volume loss based VS hemoglobin concentration based ) based blood transfusion practices in patients undergoing major oncological surgery for pelvic or spinal tumor and investigate their postoperative complications.

DETAILED DESCRIPTION:
260 patients underwent major oncological surgery for open pelvic or spinal tumor resection were included in this study. We looked at white blood cells, hemoglobin, hematocrit, neutrophil ratio, C-reactive protein, erythrocyte sedimentation rate, and IL-6 levels 1 day, 3 days, and 7 days after surgery The main question it sought to answer was whether there was a difference in postoperative complications 30 days after surgery between patients who received blood transfusions based on volume loss and those who received blood transfusions based on hemoglobin concentration during surgery.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 70
* patients with pelvic or spinal tumor
* conduct open resection surgery for tumor removal
* with expected surgery duration greater than 3 hours
* with expected blood loss greater than 400 ml

Exclusion Criteria:

* age < 18 or >70
* Limb tumor patients or patients with pelvic and spinal tumors undergoing closed internal fixation or vertebroplasty or minimally invasive surgery
* received chemotherapy or immunotherapy before surgery
* with expected surgery length less than 3 hours
* with expected intraoperative blood loss less than 400ml

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
percentage of the postoperative complication | patients were carefully followed for complication occurrence 1 month after surgery.
  Major postoperative complications include but are not limited to surgical site infection, lung infection, deep vein thrombosis, pressure ulcers and so on

SECONDARY OUTCOMES:
transfusion of red packed blood cells | during hospitalization after surgery, an averagy of 1 week
  total volume of blood transfusion calculated after surgery
length of hospital stay | during hospitalization after surgery, an averagy of 1 week
  Number of days patients stay in hospital after surgery.
White blood cell count | 1 day，3 days，7 days，and 30 days after surgery
  White blood cell count was measured in patients 1 day, 3 days, and 7 days and 30 days after surgery.
hemoglobin level | 1 day，3 days，7 days，and 30 days after surgery
  hemoglobin level was measured in patients 1 day, 3 days, and 7 days and 30 days after surgery.
hematocrit | 1 day，3 days，7 days，and 30 days after surgery
  hematocrit was measured in patients 1 day, 3 days, and 7 days and 30 days after surgery.
neutrophil ratio | 1 day，3 days，7 days，and 30 days after surgery
  the neutrophil ratio was measured in patients 1 day, 3 days, and 7 days and 30 days after surgery.
C-reactive protein | 1 day，3 days，7 days，and 30 days after surgery
  C-reactive protein was measured in patients 1 day, 3 days, and 7 days and 30 days after surgery.
erythrocyte sedimentation rate | 1 day，3 days，7 days，and 30 days after surgery
  erythrocyte sedimentation rate was measured in patients 1 day, 3 days, and 7 days and 30 days after surgery.
nterleukin-6 level | 1 day，3 days，7 days，and 30 days after surgery
  Interleukin-6 level was measured in patients 1 day, 3 days, and 7 days and 30 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaobo Yan, MD, Principal Investigator — 2nd Affiliated Hospital Of Zhejiang University

IPD SHARING:
Plan to Share IPD: No